CLINICAL TRIAL: NCT01481194
Title: An Open-Label Phase II Study of the Safety and Efficacy of Doxorubicin and Cyclophosphamide in Combination With Bortezomib, Lenalidomide, and Dexamethasone for Treatment of Patients With Newly Diagnosed Multiple Myeloma
Brief Title: ACVDL Treatment for Patients With Newly Diagnosed Multiple Myeloma
Acronym: ACVDL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDU/VS-HKU/CTC-2011-01
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Doxorubicin; Bortezomib; Lenalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACVDL (Experimental): ACVDL is a combination of doxorubicin, cyclophosphamide, bortezomib, dexamethasone, and lenalidomide
  Interventions: Drug: Doxorubicin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Doxorubicin — 50 mg/m2 IV on day 1 of a 21-day cycle
Drug: Bortezomib — 1.3 mg/m2 IV push on days 2 and 9 of a 21-day cycle
Drug: Lenalidomide — 15 mg orally on days 1-14 of a 21-day cycle
Drug: Dexamethasone — 20 mg orally on days 2, 3, 9, and 10 of a 21-day cycle
Drug: Cyclophosphamide — 750 mg/m2 IV on day 1 of a 21-day cycle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination treatment of doxorubicin, cyclophosphamide, bortezomib, dexamethasone, and lenalidomide in newly diagnosed multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years at the time of signing informed consent.
2. Subject is diagnosed with symptomatic multiple myeloma based on the International Myeloma Working Group Diagnostic Criteria (Kyle 2009):

   * Monoclonal plasma cells in the bone marrow ≥ 10% and/or presence of a biopsy-proven plasmacytoma.
   * Monoclonal protein present in the serum and/or urine. If no monoclonal protein is detected (non-secretory disease), then ≥ 30% monoclonal bone marrow plasma cells and/or a biopsy-proven plasmacytoma is required.
   * Myeloma-related organ dysfunction
3. The myeloma disease burden must be measurable with at least one of the following criteria (Durie et al. 2006):

   * Serum M-protein ≥ 10 g/l
   * Urine M-protein ≥ 200 mg/24 h
   * Involved FLC ≥ 100 mg/l provided serum FLC ratio is abnormal
   * Bone marrow plasma cells > 30%
4. Subject has a Karnofsky performance status of ≥ 60.
5. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
6. Subject is willing and able to comply with the protocol as judged by the investigator.

Exclusion Criteria:

1. Any prior systemic therapy for multiple myeloma.
2. Other therapies such as biologic therapy and chemotherapy less than 3 months prior to screening.
3. Any prior treatment with doxorubicin or other anthracycline.
4. Concurrent or recent (less than 2 weeks prior to Screening) radiotherapy or surgery.
5. Prior glucocorticoid treatment of multiple myeloma exceeding dexamethasone 20mg/day for a maximum of 7 days. Topical glucocorticosteroid therapy to treat non-malignant comorbid disorders is permitted.
6. More than or equal to grade 2 peripheral neuropathy according to the NCI-CTC criteria on clinical examination within 14 days before enrolment (Day 1 of Cycle 1).
7. Evidence of mucosal or internal bleeding and/or platelet counts < 50 x 10^9/l. Platelet transfusions may not be used to meet PLT eligibility criteria.
8. Absolute neutrophil count (ANC) < 1 x 10^9/l. Growth factors may not be used to meet ANC eligibility criteria.
9. Hemoglobin < 5.0 mmol/l. The subject may be included after correction of the hemoglobin level by transfusion or treatment with erythropoietin.
10. Alanine aminotransferase (ALAT) > 2 x ULN.
11. Myocardial infarction within 6 months prior to enrolment or New York Heart Association (NYHA) Class IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
12. Clinically relevant active infection or serious co-morbid medical conditions, such as chronic obstructive or chronic restrictive pulmonary disease, and cirrhosis.
13. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
14. Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, or in situ prostate cancer for which the subject has been disease-free for at least 3 years.
15. Female subject is pregnant or breast-feeding. The first serum pregnancy test to be done within 10-14 days prior to the study treatment start and repeated serum pregnancy test to be done within 24 hours prior to the start of study treatment.
16. Female subjects who are of childbearing potential (biologically capable of becoming pregnant) or men with partners of childbearing potential, who are unwilling or unable to use effective means of contraception. The means of contraception must be TWO acceptable methods of birth control, one highly effective method (hormonal contraceptives pills, injections or implants, tubal ligation, partner's vasectomy) and one additional effective method (condom, diaphragm, cervical cap) AT THE SAME TIME, at least 28 days before she or he starts ACVDL and for at least 28 days after the last dose of ACVDL.
17. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
18. Uncontrolled diabetes mellitus at the discretion of the investigator.
19. Hypersensitivity and/or contraindication to any one of the Investigational Medicinal Products (IMP), acyclovir or similar anti-viral drug.
20. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
21. Known HIV infection.
22. Known active hepatitis B or C viral infection.
23. Known intolerance to steroid therapy.
24. Current or recent (within 30 days prior to Screening) treatment with another investigational drug.
25. Unable to comply with the administration of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Response rate | 4 weeks after completion of 8 treatment cycles

SECONDARY OUTCOMES:
Complete response rate | 4 weeks after completion of 8 treatment cycles
Very good partial response rate | 4 weeks after completion of 8 treatment cycles
Time to progression | 4 years
Progression free survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Torben Plesner, DMSc, Study Chair — Vejle Hospital
Locations (1):
- Department of Hematology, Vejle, Denmark